CLINICAL TRIAL: NCT03461679
Title: A Randomised Controlled Trial Investigating the Addition of an Adductor Canal Block to a Femoral Triangle Block for Analgesia After Total Knee Replacement
Brief Title: Analgesic Effect of Adding an Adductor Canal Block to a Femoral Triangle Block for Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/ 2809 CGH
Record Dates: First submitted 2018-02-25; First posted 2018-03-12 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Total Knee Replacements

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Adductor canal block Femoral triangle block
  Interventions: Procedure: Adductor canal block; Procedure: Femoral triangle block
- Standard (Active Comparator): Femoral triangle block
  Interventions: Procedure: Femoral triangle block

INTERVENTIONS:
Procedure: Adductor canal block — Single shot block with 0.5% bupivacaine 10mls
  Arms: Intervention
Procedure: Femoral triangle block — Single shot block with 0.5% bupivacaine 10mls

SUMMARY:
The aim of the study is to investigate whether the addition of an adductor canal block to a femoral triangle block will provide better analgesia for patients after total knee replacements.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee arthroplasty under spinal anaesthesia
* 45y or older
* ASA 1-3
* BMI 18-35

Exclusion Criteria:

* Unable to consent
* Chronic opioid consumption
* Allergy to study medication
* Lower limb surgery preceding year
* Unable to complete baseline testing, pre-existing neurological deficit
* Contraindication to spinal anaesthesia

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours
  Morphine
Opioid consumption | 48 hours
  Morphine

SECONDARY OUTCOMES:
Muscle strength | 24 hours
  measured with dynanometer
Muscle strength | 48 hours
  measured with dynanometer
Time to up and go test | 24 hours
  Time to get up from chair, walk 3 meters and return to chair
Time to up and go test | 48 hours
  Time to get up from chair, walk 3 meters and return to chair
30 Chair stand test | 24 hours
  Number of times a patient can stand up from sitting position in 30 seconds
30 Chair stand test | 48 hours
  Number of times a patient can stand up from sitting position in 30 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No